CLINICAL TRIAL: NCT02709434
Title: The Efficacy of a Structured Psychoeducational Inflammatory Bowel Disease Group on the Control of Fatigue in an Adult Outpatient Setting for Patients With Objectively Quiescent Disease.
Brief Title: Fatigue Management in Quiescent IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LW Fatigue study
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Fatigue; Inflammatory Bowel Disease
MeSH Terms: conditions — Fatigue; Inflammatory Bowel Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Patients with quiescent IBD who are randomized to receive the active intervention of the psychoeducational programme
  Interventions: Behavioral: Psychoeducational programme; Other: Standard care
- Control group (Placebo Comparator): Randomized to standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Behavioral: Psychoeducational programme — Activity diary analysis and a structured programme of intervention
  Arms: Intervention group
Other: Standard care — Usual IBD management

SUMMARY:
Fatigue is a very frequently reported symptom in patients with inflammatory bowel disease (IBD), whether it is Crohn's disease (CD) or ulcerative colitis (UC). Sometimes the fatigue may be easily explained by other symptoms or tests which show that the disease is active. For example patients may be anaemic (have a low blood count) which can in itself lead to a feeling of being tired all the time. Treatment of the disease can make some of these patients feel less fatigued.

However, 4 or 5 out of every 10 patients with IBD which is felt to be in remission (ie not active disease) report fatigue. This can have far-reaching implications for patients in their everyday lives, with issues around work or school, close relationships, travel and leisure being profoundly affected. The CCUK funded research on fatigue and IBD, led by Professor Christine Norton and Wladzia Czuber-Dochan at King's College London, has identified fatigue as being a significant issue facing patients and has also highlighted that few doctors offer help and support beyond treating the disease itself when active. This is partly because fatigue itself has been difficult to measure and so any study designed to treat fatigue would be limited by being unable to quantify any improvement in a meaningful way.

Fortunately the King's College group have developed a 'fatigue score' which is a simple questionnaire that is able to quantify the severity of fatigue. The aim of our study is to assess the effect of a structured support and educational programme on the levels of fatigue in patients with inactive IBD who report moderate or severe levels of fatigue. A secondary component of our study is to see if there are any associations between fatigue levels and disease activity or other parameters such as quality of life, anxiety or symptoms of overlapping irritable bowel syndrome.

Patients will be approached in the out-patient or telephone clinics and the study will be explained with written information and any questions will be answered. If they agree to being involved they will be asked to complete the fatigue and a number of other questionnaires in addition to having the standard assessment of symptoms, blood tests and a stool specimen. Patients with active disease will be excluded from the subsequent group interventions but the data they have provided to this point will still be helpful in our understanding of fatigue in IBD. Patients identified as being in remission following the initial assessments will be offered the opportunity to be involved in the next stage of the study. The stool samples will also be analysed for the microbiome ie which bacteria are present as some studies suggest that patients with IBD may have a reduced diversity of bacteria in their intestines.

Half of this group will be randomised to active intervention and half will act as a control group for the rest of the study. The active intervention will involve completion of activity diaries over the following two weeks and then analysis of the diaries and agreement on behaviour changes designed to help fatigue. This will be supported by written information and three, monthly small group sessions to reinforce and support these changes.

At the end of the study all patients will again complete the fatigue and quality of life questionnaires and have their disease activity assessed by symptom scores, blood and stool tests. The baseline results and the final results will be analysed to see if there is any improvement in fatigue in the group undergoing the programme of support and behaviour change.

This is only a small pilot study but if it demonstrates that the intervention is feasible and may help with fatigue then a larger study will be performed to try and confirm our initial findings.

Our ultimate aim is to find a simple intervention to empower patients to deal with the difficult task of living with IBD and the fatigue that this can bring.

DETAILED DESCRIPTION:
Background

41%- 48% of patients with inflammatory bowel disease (IBD), which is in remission, experience fatigue (1). Fatigue is associated with significant physical, emotional, psychological and social consequences (2). This can have wide-reaching implications for patients in their everyday lives, with issues around work productivity, academic achievement, close relationships, travel and leisure being profoundly affected. Based on data from the CCUK national lottery-funded research on fatigue, although 68% of responding IBD treating professionals felt that fatigue was adequately treatable less than half offer anything over and above checking the haemoglobin level and treat if low, with only around one third offering lifestyle related advice on diet, exercise and sleep (3). The CCUK funded research on fatigue and IBD led by Professor Christine Norton and Wladzia Czuber-Dochan has not only identified fatigue as a significant issue facing patients but has also developed an objective fatigue score to quantify it. Leading on from this the King's College team has studied the role of diet and exercise in fatigue.

Aims of the proposed investigation

Our study aims to address two key questions:

1. Do patients with active IBD have higher fatigue scores than patients with inactive disease? This question will be addressed as we will be screening a selection of patients coming to the specialist IBD clinic. Some will have active disease when assessed and so will be excluded from further interventional study. Others with inactive disease will be recruited to the study, but we will be able to compare fatigue scores in both the active and inactive disease groups. In addition we will explore any association between fatigue scores and anxiety/depression, somatisation scores, quality of life, overlapping IBS symptoms and the faecal microbiome.
2. Can the intervention of planned behavioural change improve the symptoms of fatigue in patients with inflammatory bowel disease in remission?

We believe our study complements the existing work on fatigue by offering a structured psychoeducational intervention centred around a self-management booklet and group-work. The primary outcome of the study is to assess fatigue in an IBD remission cohort. The study will be undertaken by Lisa Warren under the supervision of Dr Anthony O'Connor and Dr John Hamlin with input from Debbie Pullen (mental health nurse specialist) and Anna Errington (occupational therapist, department of liason psychiatry).

Secondary outcomes for a larger study that could cascade from this pilot would be to assess if there is a decreased risk of flare and an improved quality of life in patients in whom fatigue is adequately managed.

Detailed plan of investigation and methodology

All patients being screened for this study will be required to give informed consent. In order to recruit the proposed study numbers for the active intervention we estimate that we will have to screen approximately 100 patients. A large number of patients may be excluded from the active intervention study as baseline clinical and laboratory investigations, completed as part of their standard disease assessment, will suggest they have active disease. However data collected on these patients will still provide valuable information about fatigue in patients with IBD, such as any association between fatigue score and severity of active disease, or other parameters such as somatisation score (as assessed by PHQ15 form), quality of life (SIBDQ & SF36), overlapping IBD symptoms (Rome III criteria), or anxiety and depression (HAD score).

Patients identified as being in remission will be offered the opportunity to be involved in the psychoeducational interventional study. The study will be explained with written information and any questions will be answered. If they agree to being involved they will be asked to complete the fatigue questionnaire in addition to questionnaires addressing anxiety/depression (HAD), somatisation (PHQ15), overlapping irritable bowel syndrome symptoms (Rome III), and quality of life (SIBDQ & SF36). In addition, patients will have the standard assessment of disease activity with symptoms, blood tests, and stool specimens. The stool sample will be sent for faecal calprotectin measurement which is a non-invasive and sensitive marker of bowel inflammation. The stool samples will then also be stored for future assessment of the faecal microbiome (the different bacteria in the intestine) in order to examine any association between this and disease activity, fatigue scores, or the other parameters assessed with the questionnares.

Patients with active inflammation based on symptoms, blood tests, or stool calprotectin level will be excluded from the subsequent psychological intervention aspect of the study.

Those with inactive disease will be randomized, by concealed envelopes, in to two groups. The first group will act as the control and continue current management. The active intervention group will complete activity diaries over the following two weeks. The active intervention will be an analysis of the activity diaries and agreement on behaviour changes designed to help fatigue. This will be supported by written information and three, monthly small group sessions to reinforce and support these changes.

At the end of the study all patients will again complete the fatigue and other questionnaires outlined above and they will have their disease activity assessed by symptom scores, blood and stool tests. The baseline results and the final results will be analysed to see if there is any improvement in fatigue in the group undergoing the programme of support and behaviour change.

This is only a small pilot study but, if it demonstrates that the intervention is feasible and may help with fatigue, then a larger study will be performed to try and confirm our initial findings. Our data will also help inform IBD specialists and their patients about factors which may play a role in the common symptom of fatigue.

Our ultimate aim is to find a simple intervention to empower patients to deal with the difficult task of living with IBD and the fatigue that this can bring.

Our active intervention study group will be patients with inactive disease only, in order to avoid confounding factors. Those patients with inactive disease will all complete activity diaries and half of these will be randomised to the active intervention.

As there are no proven interventions to treat IBD-related fatigue we do not forsee ethical problems relating to the other half of patients being randomised to no intervention, other than their existing treatment.

The psychoeducational intervention of behaviour changes centred around a self-management booklet will be made by our IBD clinical nurse specialist, with support from the mental health team who are trained in these interventions.

Participants :

We plan to recruit 20 IBD patients, 10 with Ulcerative Colitis (UC) and 10 with Crohn's Disease (CD) with disease in remission for the active intervention arm and 20 IBD patients in remission for the control group. Remission for CD will be defined as Harvey-Bradshaw Index (HBI) <5 and C-reactive protein (CRP) <5. For UC it will be defined as partial Mayo score ≤2 and CRP <5. For both groups a faecal calprotectin (FC) of > 250ug/g will be regarded as indicating active disease and will exclude patients from the study. Patients will also be excluded if they are anaemic (Hb <14g/dL for males, 11.5g/dL for females). In the CD arm patients will be assessed for Vitamin B12 and Vitamin D status and excluded if B12 is less than 300 pmol/l or Vitamin D less than 30 ng/mL.

Interventions :

We intend to commence recruitment in January 2016 via our twice-weekly IBD out-patient clinics in addition to nurse-led telephone clinics. We aim to complete recruitment within 3 months with the interventions scheduled to begin in February.

At week zero the patients will be provided with information leaflets about the study and the process will be explained and questions answered. Those patients giving informed consent will be screened for baseline measurements including the CCUK fatigue score, in addition to completing the other questionnaires outlined in the methodology above. Baseline blood and stool samples will be taken to assess disease activity. Patients deemed to have active disease will be excluded from the rest of the study and their medical management optimised in line with local and national guidelines. Those patients meeting the inclusion criteria will be provided with activity diaries and asked to complete them over the following 4 weeks. All patients will have their baseline data analysed to study any association between fatigue scores and disease activity (as measured by HBI/Mayo score, CRP, FC), quality of life (as measured by SF36 & S-IBDQ), anxiety and depression (HAD) or somatisation (PHQ15).

After excluding patients with active disease we will randomise the study population into two groups. Randomisation will be by allocation from concealed envelopes by a physician not involved in the study. The nature of the study itself means that it will not be blinded. As this is a pilot study and there is no existing data on the effect of this intervention on fatigue we have not performed a power calculation for study population size. The active group will have analysis of their activity diary and agree behaviour changes. This group will have three subsequent visits taking place on a monthly basis until week 20, consisting of small group work of 4 patients per session to reinforce behaviour changes. At week 20, the patients will come for a 6th and final visit at which response will be assessed. This will involve disease assessment with clinical indices, repeat blod and stool samples and completion of the same questionnaires as baseline. The control group will have standard medical management but will also be reviewed at week 20 and undergo the same assessments.

Comparators :

Age, sex and disease matched controls will be identified from our IBD clinic.

Outcomes :

At the sixth visit (week 20) Fatigue score (and other questionnaires as outlined above), CRP, FC and HBI or partial Mayo Score will be obtained.

Timetable

Potential application of results, including benefits for people living with IBD

We feel that patients with fatigue when in remission currently do not have sufficient access to interventions designed specifically to manage fatigue as a symptom. In the CCUK fatigue study there was a clear message from professionals that they wished to have a greater array of evidence based interventions to offer patients under such circumstances. We believe our intervention, which offers supported non-pharmacologic self-management, will be empowering and worthwhile. We feel that this work would complement the sterling work undertaken by CCUK on fatigue in IBD in recent years. Interest has been expressed throughout the Yorkshire and Humber Royal College of Nursing IBD Network in using the booklet and method should it prove effective.

Dissemination intentions

We expect to publish our findings in abstract form and are hopeful that this pilot study will enable us to assess the feasibility of commencing an MSc or PhD project in facilitating group work for fatigue management in our IBD cohort. Dr Hamlin has been in conversation with Wladzia Czuber-Dochan from King's College and their group has discussed our proposal. They feel that this is an interesting project with no conflict with their existing studies. They also expressed an interest in collaborating with us on future studies should this pilot study provide some interesting preliminary data.

Key references

1. Van Langenberg DR and Gibson PR, 2010: Systematic review; fatigue in inflammatory bowel disease. Alimentary Pharmacol Therapy July 2010;32(2) 131-143
2. Gasche C et al, 2004: Iron, anaemia and inflammatory bowel disease. Gut August 2004; 53(8) 1190-1197
3. CCUK Fatigue in IBD study http://www.fatigueinibd.co.uk/research/outcomes/

ELIGIBILITY:
Inclusion Criteria:

* Patiets with IBD in clinical and biochemical remission with no other obvious identifiable explanation for their fatigue

Exclusion Criteria:

* Patients with active inflammation based on symptoms, blood tests, or stool calprotectin level will be excluded from the subsequent psychological intervention aspect of the study. Patients unable to give informed consent or who are unable to understand and follow the intervention will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Fatigue score | 20 weeks

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] O'Connor A, Ratnakumaran R, Warren L, Pullen D, Errington A, Gracie DJ, Sagar RC, Hamlin PJ, Ford AC. Randomized controlled trial: a pilot study of a psychoeducational intervention for fatigue in patients with quiescent inflammatory bowel disease. Ther Adv Chronic Dis. 2019 Mar 26;10:2040622319838439. doi: 10.1177/2040622319838439. eCollection 2019. PMID 30937156